CLINICAL TRIAL: NCT02194426
Title: A Phase I Multi-centre, Open-label, Repeated-dose, Dose-escalation Study to Assess Safety, Tolerability and Pharmacokinetics of MP0250 in Patients With Advanced Solid Tumours
Brief Title: First-in-human Study to Investigate the Safety, Tolerability and Blood Levels of the Test Drug MP0250 in Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Molecular Partners AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP0250-CP101; 2014-000366-21 (EudraCT Number)
Record Dates: First submitted 2014-06-12; First posted 2014-07-18 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2018-04

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — MP0250

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MP0250 (Experimental): see section "intervention description" below
  Interventions: Drug: MP0250

INTERVENTIONS:
Drug: MP0250 — Intravenous application by infusion of MP0250 at up to six dose levels, every other week for up to 24 infusions.

SUMMARY:
This research study is looking at a new DARPin® drug candidate, called MP0250. There is evidence from preclinical studies that MP0250 may be effective in the treatment of cancer. This is the first study of MP0250 in humans and its main purpose is to test its safety and tolerability in patients with cancer. This study will also examine how the drug is changed by and removed from the body and look for indicators that the drug may be effective against cancer. This study will test several different dose levels of the study drug to determine the safety and tolerability profile of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. Histologically confirmed and documented advanced or metastatic solid tumour refractory to at least 1 prior regimen of standard treatment or for which no curative therapy is available and for whom MP0250 is a reasonable option
3. Progressive or stable disease documented radiologically in the 4 weeks prior to screening
4. Presence of a measurable tumour or a tumour evaluable per RECIST v1.1
5. ECOG performance status ≤ 1
6. Life expectancy ≥ 12 weeks
7. Adequate haematological function prior to first dose, defined as:

   * Absolute neutrophils count ≥ 1500 cells/μL
   * Haemoglobin ≥ 9 g/dL
   * Platelet count > 100,000/μL
   * Prothrombin time or partial thromboplastin time < 1.2 x ULN
8. Adequate renal function prior to first dose, defined as either

   * Serum creatinine < 1.5 mg/dL or
   * Serum creatinine clearance ≥ 50 mL/min/m2 (by Cockroft-Gault equation)
9. Adequate hepatic function prior to first dose, defined as

   * Total bilirubin ≤ 1.5 x ULN
   * AST/ALT ≤ 2.5 x ULN, or ≤ 5 x ULN if known hepatic metastases
   * Alkaline phosphatase ≤ 2.5 x ULN, or ≤ 5 x ULN if known hepatic or bone metastases
10. Female patients with a negative pregnancy test result at screening and baseline

Exclusion Criteria:

1. Female patients pregnant or breast-feeding
2. Haematological malignancies or other secondary malignancy, that is currently clinically significant or requires active intervention
3. Known untreated or symptomatic brain metastases
4. Predominantly squamous non-small cell lung carcinoma
5. Anti-tumour treatment within 4 weeks of the first infusion of MP0250, such as chemotherapy, experimental or targeted therapy, biologics, hormonal therapy and radiotherapy. The anti-tumour treatments below need longer wash-out periods and must not be given within the indicated weeks of the first infusion of MP0250:

   i. Nitrosoureas: 6 weeks ii. Monoclonal antibodies: 8 weeks
6. Exceptions: the following anti-tumour treatments are allowed as indicated i. Palliative radiation to bone metastases to relieve bone pain ii. Standard of care treatment such as bone modifying agents (i.e. bisphosphonates), denosumab, maintenance hormonal therapy for metastatic prostate and breast cancers, hormone-replacement therapy, and oral contraceptives
7. Presence of residual toxicities of CTC-AE Grade ≥ 2 after prior anti-tumour therapy at screening. Except meeting other exclusion criteria, grade 1 toxicities related to previous treatments are acceptable at the time of the first infusion of MP0250, as well as Grade 2 alopecia
8. Exclusion criterion removed
9. Major surgical procedures, open biopsy or significant traumatic injury within 4 weeks of first dose or anticipation of major surgical procedure during the course of the study, core biopsy or minor surgical procedures within 1 week of first dose
10. Serious non-healing wound, active ulcer or untreated bone fracture
11. Proteinuria at screening as defined by ≥ 1+ on urinalysis dipstick, confirmed by ≥ 1g in 24h urinalysis
12. Uncontrolled hypertension or any other serious cardiovascular or cardiac condition as judged by the investigator
13. Severe or uncontrolled renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-07; Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with dose limiting toxicities | From the Day 0 (first infusion) up to 35 days
Vital signs | From inclusion (week -4) up to week 56
Frequency of adverse events | From inclusion up to week 56
MP0250 plasma concentration-time profile | From Day 0 (first infusion) up to week 56
Nature of dose limiting toxicities | From the Day 0 (first infusion) up to 35 days
Nature of adverse events | From inclusion up to week 56
Severity of adverse events | From inclusion up to week 56
Blood chemistry values | From inclusion (week -4) up to week 56
Haematology values | From inclusion (week -4) up to week 56
Urine values | From inclusion (week -4) up to week 56
Electrocardiogram measurements | From inclusion (week -4) up to week 56
Pharmacokinetics parameters | From Day 0 (first infusion) up to week 56

SECONDARY OUTCOMES:
Incidence of anti-drug-antibodies | From the Day 0 (first infusion) up to week 56
Titre of anti-drug-antibodies | From the Day 0 (first infusion) up to week 56

CONTACTS AND LOCATIONS:
Locations (4):
- Study Site Barcelona, Barcelona, Catalonia, Spain
- Study Site St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland
- United Kingdom (2):
  - Study Site Cambridge, Cambridge, Cambridgeshire
  - Study Site Oxford, Oxford, Oxfordshire

REFERENCES:
- [Derived] Baird RD, Linossi C, Middleton M, Lord S, Harris A, Rodon J, Zitt C, Fiedler U, Dawson KM, Leupin N, Stumpp MT, Harstrick A, Azaro A, Fischer S, Omlin A. First-in-Human Phase I Study of MP0250, a First-in-Class DARPin Drug Candidate Targeting VEGF and HGF, in Patients With Advanced Solid Tumors. J Clin Oncol. 2021 Jan 10;39(2):145-154. doi: 10.1200/JCO.20.00596. Epub 2020 Dec 10. PMID 33301375